CLINICAL TRIAL: NCT04423081
Title: Cross-cultural Adaptation and Validation of the French Version of the EXIT (EXperiences of Induction Tool) Self-questionnaire Assessing Women's Feelings About the Onset of Childbirth
Brief Title: Cross-cultural Adaptation and Validation of the French Version of the EXIT (EXperiences of Induction Tool) (EXIT)
Acronym: EXIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 GALLOT; 2020-A01286-33. (Other: ANSM)
Record Dates: First submitted 2020-05-26; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Induction of Labor
Keywords: EXIT scale; induction of labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EXIT scale — completion of EXIT scale translated in french

SUMMARY:
The objective of the study is to cross-culturally adapt and validate the French version of the EXIT scale: an assessment tool on induction of labor.

DETAILED DESCRIPTION:
Favourable agreement was obtained from the authors to adapt the Australian moose tool in a cross-cultural manner. None of the co-authors expressed a desire to collaborate on our project. The EXIT questionnaire is free of rights.

The translation of the EXIT questionnaire into French will be carried out according to the recommended steps of the cross-cultural adaptation process (21, 22, 25): translation of the source version into French by three native French translators, adaptation of the different translations by a group of experts, back translation by two native English speakers, testing with a panel of women who have been triggered for childbirth, in order to arrive at the final version which will be evaluated in a sample of the target population.

Information about the study will be given to women between Day 2 and Day 4 postpartum. Patients' non-opposition to participate in this study will be collected in the patient's medical record.

Recruitment of subjects: the study will be proposed to all eligible women who have been induced for their delivery and with an unfavourable cervix in the obstetrics department of the CHU Estaing, Clermont-Ferrand.

Completion of the questionnaire: women will complete the EXIT self-questionnaire between D2 and D4 post-delivery.

The data collection will include additional socio-demographic and clinical information for each woman participating in the study from their medical records.

The test-retest involves filling in the EXIT questionnaire twice at one to two week intervals.

The women will be contacted by phone one week after the first EXIT test, to inform them that a link will be sent by e-mail to complete the EXIT questionnaire online (on Redcap) a second time. They will be called back a second time a week later if the questionnaire is not completed online.

ELIGIBILITY:
Inclusion Criteria:

* Patients having given birth in the obstetrics department of CHU Estaing, Clermont-Ferrand
* with an induction of labor
* with an unfavorable cervix (Bishop score <6)
* on living child(ren)
* Patients aged 18 years and over, understanding, speaking and reading French
* no object to participating in the study.

Exclusion Criteria:

* Patients induced at first with syntocinon.
* Patients who do not have an internet connection and an e-mail address.
* Patients under legal protection (guardianship, tutorship).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having given birth in the obstetrics department of CHU Estaing, Clermont-Ferrand with an induction of labor and with an unfavorable cervix (Bishop score <6)
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The psychometric properties of the French version of the EXperiences of Induction Tool | Day 2
  The psychometric properties of the French version of the EXperiences of Induction Tool include: acceptability, internal structure validity, convergent validity, structure validity against external criteria and reproducibility. EXperiences of Induction Tool is composed of 3 dimensions: "Time taken to give birth", "Discomfort with IOL" and "Experience of subsequent contractions". Each dimension has a minimum score of 0 and a maximum score of 5. For the dimension "Time taken to give birth, a high score mean a more positive feeling. For "Discomfort with IOL"a high score mean more discomfort. For "Experience of subsequent contractions", a high score mean a more positive feeling.

SECONDARY OUTCOMES:
Score of the EXperiences of Induction Tool | Day 2
  Score of the EXperiences of Induction Tool will be calculated. EXperiences of Induction Tool is composed of 3 dimensions: "Time taken to give birth", "Discomfort with IOL" and "Experience of subsequent contractions". Each dimension has a minimum score of 0 and a maximum score of 5. For the dimension "Time taken to give birth, a high score mean a more positive feeling. For "Discomfort with IOL"a high score mean more discomfort. For "Experience of subsequent contractions", a high score mean a more positive feeling.
Time of birth | at birth
  delay between induction of labor and birth will be calculated
time of labor start | at birth
  delay between induction of labor and labor start will be calculated
Methods of induction of labor | at birth
  the type of strategy used for induction of labor will be recored
Maternal complications | up to 1 week
  maternal complications include intra-uterine infection, endometritis, c-section, instrumental delivery, post-partum hemorhage, episiotomy
Neonatal complications | up to 1 week
  maternal complications include Apgar score < 7 to 5min, pH and lactates on umbilical arterial sampling, 2nd line operation, and rate of transfer to Intensive care unit, maternal-fetal infection

CONTACTS AND LOCATIONS:
Overall Officials: Denis Gallot, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France